CLINICAL TRIAL: NCT06867991
Title: Safety and Efficacy of Combined B Cell Depleting theRapy And Daratumumab In Autoimmune Encephalitis
Acronym: RADIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADIA-2024-11
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Anti-N-Methyl-D-Aspartate Receptor Encephalitis
Keywords: Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Ofatumumab; Daratumumab; severe autoimmune encephalitis
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Autoimmune Diseases of the Nervous System | interventions — daratumumab; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- B cell depleting agent（ofatumumab）combined with daratumumab treatment group (Experimental): The group receiving B cell depletion plus daratumumab will receive daratumumab intravenously (on the second day of ofatumumab) in addition to ofatumumab, with a dose of 8 mg/kg at weeks 0, 1, 2, and 4, and a dose of 4 mg/kg at weeks 8, 12, 16, 20, and 24. The study will investigate the effect of up to 24 cycles of daratumumab
  Interventions: Drug: Ofatumumab combined with daratumumab
- Ofatumumab treatment group (Active Comparator): Ofatumumab group received subcutaneous injection of ofatumumab at weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24
  Interventions: Drug: Ofatumumab
- Repeated intravenous immunoglobulin/plasma exchange therapy group (Active Comparator): At least two cycles of intravenous immunoglobulin/plasma exchange therapy
  Interventions: Drug: Repeated intravenous immunoglobulin/plasma exchange therapy

INTERVENTIONS:
Drug: Ofatumumab combined with daratumumab — All participants will begin acute first-line therapy prior to randomization, and participants who were receiving oral or intravenous corticosteroids at baseline will need to taper their doses according to a standard taper schedule starting 4 weeks after randomization (week 4). Patients will be randomly assigned to receive ofatumumab followed by daratumumab or ofatumumab followed by repeated intravenous globulin. The ofatumumab group will receive subcutaneous ofatumumab at weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24, while the ofatumumab-daratumumab group will receive daratumumab intravenously (on the second day of ofatumumab) in addition to ofatumumab, with a dose of 8 mg/kg at weeks 0, 1, 2, and 4, and a dose of 4 mg/kg at weeks 8, 12, 16, 20, and 24. The study will investigate the effects of up to 24 cycles of daratumumab.
  Arms: B cell depleting agent（ofatumumab）combined with daratumumab treatment group
Drug: Ofatumumab — All participants were started on acute first-line therapy before randomization, and participants who were receiving oral or intravenous glucocorticoids at baseline were required to taper their doses according to a standard taper schedule starting 4 weeks after randomization (week 4). Ofatumumab was administered subcutaneously at weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24 in the ofatumumab group.
  Arms: Ofatumumab treatment group
Drug: Repeated intravenous immunoglobulin/plasma exchange therapy — Repeated intravenous immunoglobulin/plasma exchange therapy
  Arms: Repeated intravenous immunoglobulin/plasma exchange therapy group

SUMMARY:
Autoimmune encephalitis is an autoimmune disease of the central nervous system that targets neuronal autoantigens. Anti-neuronal autoantibodies are produced in patients, with anti-NMDAR antibody being the most common.Anti-NMDAR encephalitis can be severe and life-threatening. Anti-NMDAR autoantibodies against neurons are pathogenic and are mainly produced by autoreactive B cells and plasma cells. Therefore, early elimination of these abnormal immune cells is crucial for rapid improvement of the patient's condition. This study aims to explore the efficacy and safety of B cell depletion therapy (ofatumumab) followed by plasma cell depletion therapy (daratumumab) in the treatment of severe anti-NMDAR autoimmune encephalitis.

DETAILED DESCRIPTION:
Autoimmune encephalitis (AE) is a broad spectrum of immune-mediated neuropsychiatric diseases, usually associated with antibodies against surface proteins, ion channels, synapses or intracellular proteins of neuronal cells. Anti-N-methyl-D-aspartate receptro (NMDAR) encephalitis is the most common type of AE.The clinical manifestations include behavioral changes, psychiatric symptoms, epileptic seizures, memory and cognitive deficits, abnormal movements, autonomic dysfunction and decreased consciousness. Most children and adult patients present with a syndrome that combines the above symptoms and can be severe.

Early initiation of immunotherapy is necessary to improve clinical prognosis and reduce its recurrence.

However, no disease-modifying therapy specifically for AE has been approved. A variety of therapies have emerged for severe autoimmune encephalitis, including anti-CD20 monoclonal antibody rituximab, proteasome inhibitor bortezomib, anti-CD38 monoclonal antibody daratumumab, anti-IL-6R monoclonal antibody tocilizumab, low-dose IL-2, and intrathecal methotrexate. The evidence for the efficacy of these drugs mostly comes from case reports, and there are currently no high-quality randomized controlled clinical studies reported.

Studies have found that anti-NMDAR antibody is produced by autoreactive B cells and plasma cells. Among these cells, long-lived plasma cells in the intrathecal, meningeal, and brain parenchyma are responsible for the production of pathogenic antibodies in severe cases. The B cell-depleting therapeutic antibody rituximab targets CD20-positive B cells. CD138-positive plasma cells lack CD20 surface receptors, are not targeted by rituximab, and are also resistant to other immunosuppressive therapies. Daratumumab is an anti-CD38 antibody that can target long-lived plasma cells and has shown good therapeutic responses in autoimmune hemolytic anemia, systemic lupus erythematosus, and autoimmune encephalitis, with an acceptable safety profile. Daratumumab not only works by clearing plasma cells, but also regulates certain T cell functions.

RADIA study is an investigator-initiated, randomized, controlled, open-label, multicenter clinical trial to investigate the safety and efficacy of anti-CD20 mAb ofatumumab in combination of anti-CD38 mAb daratumumab in patients with severe anti-NMDAR encephalitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 years and above
2. Meet the diagnosis of autoimmune encephalitis and the target antigen is a neuronal surface antigen
3. Have received at least 3 days of 500-1000mg high-dose methylprednisolone impulse treatment and IVIG (0.4g/kg/d for 5 consecutive days) or at least 5 plasma exchange/immunoadsorption or at least 2 times of efgartigimod treatment
4. mRS ≥ 3 points and neuropsychiatric manifestations inadequate to symptomatic treatment
5. Informed consent or guardian signed informed consent

Exclusion Criteria:

1. Severe active or chronic infection in the opinion of the investigator.
2. Concurrently/previously participated in another clinical study involving investigational therapy within 4 weeks or 5 published half-lives of the investigational therapy (whichever is longer) before randomization.
3. Women who are lactating or pregnant, or intend to become pregnant at any time within six months from study enrollment to the last dose of study drug.
4. Known history of allergy or reaction to any component of the investigational drug formulation, or history of allergic reaction after any biological treatment.
5. Any of the following at screening (one repeat test may be performed during the same screening period to confirm results prior to randomization):

   Aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN)

   Alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN)

   Total bilirubin > 1.5 × ULN (unless due to Gilbert's syndrome)

   Platelet count < 75,000/μL (or < 75 × 109/L)

   Hemoglobin < 8 g/dL (or < 80 g/L)

   Total white blood cell count < 2,500 cells/mm3

   Total immunoglobulins < 600 mg/dL

   Absolute neutrophil count < 1200 cells/μL

   CD4 T lymphocyte count < 300 cells/µL

   Receipt of any experimental B cell depleting agent, unless CD19 B Cell levels have returned to above the lower limit of normal before randomization A history of severe drug allergies or anaphylaxis to two or more foods or drugs (including known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamines, and methylprednisolone or equivalent glucocorticoids).

   A known history of primary immunodeficiency (congenital or acquired) or underlying conditions, such as human immunodeficiency virus (HIV) infection or splenectomy, that predispose the participant to infection.

   Any of the following received within 3 months before randomization Natalizumab (Tysabri®) Cyclosporin Methotrexate Mitoxantrone Cyclophosphamide Azathioprine
6. Confirmed positive hepatitis B serology (hepatitis B surface antigen and core antigen) and/or positive hepatitis C PCR at screening.
7. History of cancer, other than ovarian or extraovarian teratoma (also known as dermoid cyst) or germ cell tumor, or cutaneous squamous cell carcinoma or cutaneous basal cell carcinoma. Treatment of squamous cell carcinoma and basal cell carcinoma should have documented successful curative treatment more than 3 months before randomization.
8. Received any live or attenuated vaccine (inactivated vaccine is acceptable) within 3 weeks before enrollment.
9. Received BCG vaccine within 1 year before enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Time to mRS<=2, i.e. the proportion of patients with mRS scores of 0-2 | week 16
  Primary objective:
  • Patients achieve good outcome
  Primary endpoint:
  • Time to mRS<=2, i.e. the proportion of patients with mRS scores of 0-2

SECONDARY OUTCOMES:
mRS score at 16 weeks | After 16 weeks of treatment
  mRS score at 16 weeks
CASE score at 16 weeks | After 16 weeks of treatment
  CASE score at 16 weeks
Incidence of adverse events | After 48 weeks of treatment
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided